CLINICAL TRIAL: NCT01576055
Title: Evaluation of the GORE TIGRIS Vascular Stent in the Treatment of Atherosclerotic Lesions of the Superficial Femoral and Proximal Popliteal Arteries
Brief Title: Evaluation of the GORE TIGRIS Vascular Stent
Acronym: TIGRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCE 09-02
Record Dates: First submitted 2012-03-29; First posted 2012-04-12 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-09

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Superficial Femoral Artery; Proximal Popliteal Artery; PAD; SFA; PPA; Stent; Gore; Bare Metal Stent; LifeStent; atherosclerosis; Heparin; claudication; leg pain
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TIGRIS Vascular Stent (Experimental): GORE TIGRIS Vascular Stent
  Interventions: Device: TIGRIS Vascular Stent
- BARD LifeStent (Active Comparator): BARD LifeStent
  Interventions: Device: BARD LifeStent

INTERVENTIONS:
Device: TIGRIS Vascular Stent — Implant
  Arms: TIGRIS Vascular Stent
Device: BARD LifeStent — Implant
  Arms: BARD LifeStent

SUMMARY:
The primary objective of the randomized study is to evaluate the safety and effectiveness of the TIGRIS Vascular Stent in the treatment of de novo and restenotic atherosclerotic lesions, ≤ 24cm in length, in the superficial femoral and proximal popliteal arteries (SFA/PPA) of patients with symptomatic peripheral arterial disease (PAD).

ELIGIBILITY:
Inclusion Criteria:

* Rutherford Class 2 - 4.
* Abnormal ankle brachial index (ABI ≤0.9).
* At least 21 years of age.
* Reasonable expectation of survival of at least 12 months after the procedure.
* Male, infertile female, or female practicing an effective method of preventing pregnancy.
* One de novo or restenotic lesion of the SFA/PPA with a cumulative length visually estimated to be ≤24cm
* Arteries with reference vessel diameter of 4.0 - 6.5 mm within the SFA/PPA, estimated visually.
* Angiographic evidence of at least one patent tibial artery (<50% stenosis angiographically).
* Guidewire has successfully traversed the lesion to be treated and is within the true lumen of the distal vessel.
* Lesion has been pre-dilated before stent deployment.

Exclusion Criteria:

* Prior enrollment in this study.
* Vascular access/catheterization in the target leg within 30 days of study enrollment.
* Prior treatment of the SFA/PPA in the target leg with stenting or bypass.
* Flow-limiting aortoiliac disease.
* Additional ipsilateral femoropopliteal or tibial disease, outside of the lesion to be stented, requiring intervention.
* Arterial aneurysm in the target leg.
* Co-morbid conditions which would preclude compliance with study protocol.
* Obstructive or occlusive non-atherosclerotic disease.
* Creatinine greater than 2.5 mg/dl.
* Amputation above the metatarsals, resulting from vascular disease, in the target leg.
* Septicemia or uncontrolled infection.
* Contraindication to anticoagulation or antiplatelet therapy, including allergy to heparin, or history of heparin induced thrombocytopenia (HIT), or a positive platelet factor 4 (PF4) antibody assay.
* Abnormal platelet levels, i.e., platelet count at Baseline less than 80,000/microliter.
* History of coagulopathy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2012-04; Primary Completion 2015-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Laird, MD, Principal Investigator — UC Davis
Locations (34):
- United States (34):
  - Cardiology Associates of Mobile, Mobile, Alabama
  - Arkansas Heart, Little Rock, Arkansas
  - North County Radiology, Oceanside, California
  - UC Davis Vascular Center, Sacramento, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - First Coast Cardiovascular Institute, P.A, Jacksonville, Florida
  - MediQuest Research at Munroe Regional, Ocala, Florida
  - Orlando Regional Healthcare System, Orlando, Florida
  - Coastal Vascular & Interventional, Pensacola, Florida
  - Vascular Surgical Associates, PC, Austell, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Kaiser Permanente - Honolulu, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Alexian Brothers Specialty Group, Elk Grove Village, Illinois
  - Heart Care Research Foundation, Mokena, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - HeartCare MidWest - Peoria, Peoria, Illinois
  - Indiana University Vascular Surgery, Indianapolis, Indiana
  - Genesis Medical Center, Davenport, Iowa
  - University of Iowa, Iowa City, Iowa
  - Minneapolis Radiology and Vascular, Minneapolis, Minnesota
  - SSM Health Care, Saint Charles, Missouri
  - Vascular Research Institute, Morristown, New Jersey
  - Ohio Health Research Institute, Columbus, Ohio
  - Providence Heat & Vascular Institute, Portland, Oregon
  - Heritage Valley Health System, Beaver, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - North Central Heart Institute, Ltd., Sioux Falls, South Dakota
  - Baylor Research Institute, Dallas, Texas
  - Presbyterian Hospital, Dallas, Dallas, Texas
  - CAMC Health Education and Research Institute, Inc., Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TIGRIS Vascular Stent | BARD LifeStent
Started | 197 | 70
Completed | 178 | 64
Not Completed | 19 | 6

BASELINE CHARACTERISTICS:
Population: Per Protocol Population
Groups:
- Total: Total of all reporting groups
Arm/Group | TIGRIS Vascular Stent | BARD LifeStent | Total
Number analyzed (Participants) | 197 | 70 | 267
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (9.30) | 67.9 (8.87) | 67.0 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 21 | 77
  Male | 141 | 49 | 190
Region of Enrollment [Number; unit: participants]
  United States | 142 | 54 | 196
  Europe | 55 | 16 | 71

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint - Number of Participants Free From Major Adverse Events at 30 Days
Description: Defined as any adverse event (occurring within 30 days of the initial procedure) that causes death, target vessel revascularization (TVR), and amputation above the metatarsals in the treated leg (index limb amputation).
Time Frame: 30 Days
Population: Per Protocol Population (Participants Available for 30-Day Follow-Up)
Measure: Number; unit: participants
Arm/Group | TIGRIS Vascular Stent | BARD LifeStent
Number analyzed (Participants) | 188 | 69
participants | 187 | 69

2. Primary Outcome: Primary Efficacy Endpoint - Number of Participants With Primary Patency at 12 Months
Description: Primary patency is defined by a Peak Systolic Velocity Ratio (PSVR) ≤2.5 without target lesion revascularization (TLR) at 12 months after implantation.
Time Frame: 12 Months
Population: Per Protocol Population (Participants Available for 12-Month Follow-Up)
Measure: Number; unit: participants
Arm/Group | TIGRIS Vascular Stent | BARD LifeStent
Number analyzed (Participants) | 170 | 64
participants | 97 | 35

3. Secondary Outcome: Number of Participants With Procedural Success
Description: Successful device implantation with a residual stenosis <30% without acute (within 48 hours) serious adverse events.
Time Frame: Within 48 hours of initial device implant
Population: Per Protocol Population
Measure: Number; unit: participants
Arm/Group | TIGRIS Vascular Stent | BARD LifeStent
Number analyzed (Participants) | 197 | 70
participants | 196 | 68

4. Secondary Outcome: Number of Participants With Device Success
Description: Successful delivery of stent to the intended site and successful stent deployment.
Time Frame: Immediately following initial device implant (usually within a few minutes to an hour).
Population: Per Protocol Population
Measure: Number; unit: participants
Arm/Group | TIGRIS Vascular Stent | BARD LifeStent
Number analyzed (Participants) | 197 | 70
participants | 196 | 70

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the study initiation to submission (approximately 3 years, 4 months).
Arm/Group | TIGRIS Vascular Stent | BARD LifeStent
Serious Adverse Events (participants affected / at risk) | 102/197 | 34/70
Other Adverse Events (participants affected / at risk) | 46/197 | 18/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIGRIS Vascular Stent (N=197) | BARD LifeStent (N=70)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 5 | 2
Angina pectoris (Cardiac disorders) | 5 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 1
Cardiac arrest (Cardiac disorders) | 3 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 3 | 3
Coronary artery disease (Cardiac disorders) | 4 | 1
Coronary artery stenosis (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 4 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Retinal artery embolism (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diaphragmatic hernia (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Adverse drug reaction (General disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Device breakage (General disorders) | 0 | 1
Device dislocation (General disorders) | 0 | 1
Device occlusion (General disorders) | 3 | 1
Medical device complication (General disorders) | 1 | 0
Medical device entrapment (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Vascular stent restenosis (General disorders) | 24 | 9
Vascular stent thrombosis (General disorders) | 1 | 0
Vessel puncture site haematoma (General disorders) | 1 | 0
Vessel puncture site haemorrhage (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 2
Postoperative wound infection (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Arterial restenosis (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 2 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 1
Prescribed overdose (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 6 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain stem ischaemia (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 3 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 2
Embolic stroke (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Femoral artery dissection (Vascular disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 2 | 0
Hypertensive crisis (Vascular disorders) | 2 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 6 | 3
Peripheral arterial occlusive disease (Vascular disorders) | 4 | 2
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 16 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 1
Vessel perforation (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TIGRIS Vascular Stent (N=197) | BARD LifeStent (N=70)
Vascular stent restenosis (General disorders) | 22 | 6
Intermittent claudication (Vascular disorders) | 22 | 9
Peripheral artery stenosis (Vascular disorders) | 11 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less